CLINICAL TRIAL: NCT00524771
Title: Transatlantic Active Surveillance on Cardiovascular Safety of NuvaRing (TASC)
Acronym: TASC
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Organon (Industry)
Responsible Party: Principal Investigator, Juergen Dinger, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2007_03
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-03

CONDITIONS: Contraception
Keywords: Contraception; Contraceptive Vaginal Ring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Users of NuvaRing
- 2: Users of combined oral contraceptives

SUMMARY:
The objective of this study is to characterize and compare the risks of short- and long-term use of NuvaRing® with marketed combined oral contraceptives.

DETAILED DESCRIPTION:
This is a large, multinational, controlled, prospective, active surveillance study of women who are prescribed NuvaRing® or an oral contraceptive (OC). The study follows two cohorts. The cohorts consist of new users (starters and switchers) of two different groups of hormonal contraceptives:

* NuvaRing®
* marketed combined OCs (combined oral contraceptives)

NuvaRing® is a transparent and flexible contraceptive vaginal ring containing etonogestrel and ethinylestradiol (EE). The ring releases 15 mcg EE and 120 mcg etonogestrel daily. After insertion it remains in the upper part of the vagina for 21 days, followed by 7 ring-free days before a new ring is inserted.

The primary objective of this study is to characterize and compare the risks of short- and long-term use of NuvaRing® with marketed combined OCs. The main clinical outcomes of interest for the short and long-term follow-up are:

* Deep Venous Thrombosis (DVT)
* Pulmonary Embolism (PE)
* Acute Myocardial Infarction (AMI)
* Cerebrovascular Accidents (CVA)

Secondary objectives are:

* to analyze the drug utilization pattern of NuvaRing® and marketed OCs in a study population that is representative for typical use of the individual contraceptive methods under routine medical conditions
* to characterize the baseline risk of users of the individual formulations
* to assess the compliance of NuvaRing® users and users of marketed OCs
* to analyze the reasons for discontinuing the treatment with NuvaRing® and/or marketed OCs.

The study will use a non-interference approach to provide standardized, comprehensive, reliable information on these treatments in a routine clinical practice setting.

Study participants will be recruited via an international network of more than 1000 gynecologists. After study entry cohort members will be followed for a period of 30 to 48 months for rare serious safety outcomes. Regular, active contacts with the cohort members by the study team of the Berlin Center for Epidemiology and Health Research (ZEG), Germany will provide the necessary information on health-related events or changes in health status (= active surveillance).

Approximately 15,000 subjects per cohort will be recruited by participating physicians in order to provide approx. 86,000 women-years (WY) of observation. Subjects will be considered for enrollment in this study after the participating physician has determined that NuvaRing® or OC use is appropriate. There will be no specific inclusion/exclusion criteria. All women who are eligible are to be asked by their physician if they are willing to participate. As this a non-interventional study, the possibility to participate in the study should not be discussed with the patient before both - physician and patient - agree upon the prescription.

The study will be conducted in several European countries and the United States.

The study will be divided into 2 phases: a baseline survey which includes an initial consultation at baseline with a participating physician, and a follow-up phase which includes two follow-up contacts within the first year and then annual follow-up contacts for up to 4 years post-baseline.

The study will maintain scientific independence and will be governed by an independent Safety Monitoring and Advisory Council (SMAC). The Berlin Center for Epidemiology and Health Research (ZEG) and its research team will be accountable to the council in all scientific matters. The members of the council will be international experts in relevant scientific fields (e. g., epidemiology, drug safety, gynecology, cardiology, statistics, endocrinology).

ELIGIBILITY:
Inclusion Criteria:

* women who are prescribed NuvaRing® or a combined oral contraceptive and who are new users (Starters, restarters or switchers) of the formulation

Exclusion Criteria:

* women who do not consent to participate in the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women prescribed hormonal contraceptives by gynecologists
Sampling Method: Non-Probability Sample
Enrollment: 34100 (Actual)
Dates: Start 2007-09; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen C Dinger, MD, PhD, Principal Investigator — Center for Epidemiology and Health Research Berlin, Germany
Locations (1):
- Berlin Center for Epidemiology and Health Research, Berlin, State of Berlin, Germany

REFERENCES:
- [Result] Dinger J, Mohner S, Heinemann K. Cardiovascular risk associated with the use of an etonogestrel-containing vaginal ring. Obstet Gynecol. 2013 Oct;122(4):800-808. doi: 10.1097/AOG.0b013e3182a5ec6b. PMID 24084537

RESULTS

PARTICIPANT FLOW:
Groups:
- NuvaRing: Users of an etonogestrel-containing and ethinylestradiol-containing vaginal ring
- Combined Oral Contraceptives (COC): Users of combined oral contraceptive pills
Period: Overall Study
Arm/Group | NuvaRing | Combined Oral Contraceptives (COC)
Started | 17084 | 17016
Completed | 16864 (Numbers completed refer to first follow-up. Individual follow-up ranged between 0.5 and 4.0 years.) | 16431 (Numbers completed refer to first follow-up. Individual follow-up ranged between 0.5 and 4.0 years.)
Not Completed | 220 | 585
Not completed — Protocol Violation | 220 | 585

BASELINE CHARACTERISTICS:
Population: All study participants that were not excluded due to protocol violations.
Groups:
- Total: Total of all reporting groups
Arm/Group | NuvaRing | Combined Oral Contraceptives (COC) | Total
Number analyzed (Participants) | 16864 | 16431 | 33295
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (7.3) | 26.9 (7.6) | 27.4 (7.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 127 | 406 | 533
  Between 18 and 65 years | 16737 | 16025 | 32762
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16864 | 16431 | 33295
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Europe | 8215 | 7699 | 15914
  United States | 8649 | 8732 | 17381

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Venous Thromboembolism (VTE)
Description: Venous thromboembolism (VTE) associated with the use of hormonal contraceptives that contain both an estrogen and progestin.
Time Frame: Time to event analysis within 48 months
Population: Study participants that were not excluded due to protocol violations.
Measure: Number; unit: participants
Groups:
- COC2: A priori defined subgroup of users of combined oral contraceptive pills without desogestrel or gestodene
Arm/Group | NuvaRing | Combined Oral Contraceptives (COC) | COC2
Number analyzed (Participants) | 16864 | 16431 | 13811
participants | 19 | 26 | 21
Statistical Analysis 1: Comparison: NuvaRing vs Combined Oral Contraceptives (COC); Tested null hypothesis: VTE hazard ratio for NuvaRing vs. COCs is higher or equal to 2. This analysis represents the a priori defined primary statistical analysis; Test type: Non-Inferiority or Equivalence — Sample size calculations were based on a non-inferiority test of two exponential survival curves . These calculations are based on the following assumptions: 1) one-sided α of 0.025; 2) power (1-β) of 0.80; VTE incidence rate of 9.1 VTE/10.000 WY and 4) non-inferiority limit on hazard ratio of 2; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.5 to 1.5] — Hazard ratio was adjusted age, BMI, duration of current use and family history of VTE
Statistical Analysis 2: Comparison: NuvaRing vs COC2; Tested null hypothesis: VTE hazard ratio for NuvaRing vs. COC2 is higher or equal to 2; Test type: Non-Inferiority or Equivalence — Sample size calculations were based on the primary statistical analysis (see above); Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.4 to 1.7] — Hazard ratio was adjusted age, BMI, duration of current use and family history of VTE
Statistical Analysis 3: Comparison: NuvaRing vs Combined Oral Contraceptives (COC); Like analysis 1 (see above) but restricted to exposure period of less than 6 months; Test type: Non-Inferiority or Equivalence — Sample size calculations were based on the primary statistical analysis (see above); Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.3 to 2.2] — Hazard ratio was adjusted age, BMI, duration of current use and family history of VTE
Statistical Analysis 4: Comparison: NuvaRing vs Combined Oral Contraceptives (COC); Like analysis 1 (see above) but restricted to exposure period of 6 - 12 months; Test type: Non-Inferiority or Equivalence — Sample size calculations were based on the primary statistical analysis (see above); Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.3 to 2.6] — Hazard ratio was adjusted age, BMI, duration of current use and family history of VTE
Statistical Analysis 5: Comparison: NuvaRing vs Combined Oral Contraceptives (COC); Like analysis 1 (see above) but restricted to exposure period of > 12 months; Test type: Non-Inferiority or Equivalence — Sample size calculations were based on the primary statistical analysis (see above); Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.3 to 2.3] — Hazard ratio was adjusted age, BMI, duration of current use and family history of VTE

2. Primary Outcome: Number of Participants With Arterial Thromboembolism (ATE)
Description: Arterial Thromboembolism (ATE) associated with the use of hormonal contraceptives that contain both an estrogen and progestin.
Time Frame: Time to event analysis within 48 months
Measure: Number; unit: participants
Arm/Group | NuvaRing | Combined Oral Contraceptives (COC) | COC2
Number analyzed (Participants) | 16864 | 16431 | 13811
participants | 5 | 8 | 6
Statistical Analysis 1: Comparison: NuvaRing vs Combined Oral Contraceptives (COC); Test type: Non-Inferiority or Equivalence — Sample size calculations were based on the primary statistical analysis (see above); Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.2 to 2.3] — The hazard ratio was adjusted for age, BMI, Smoking, and treated hypertension
Statistical Analysis 2: Comparison: NuvaRing vs COC2; Test type: Non-Inferiority or Equivalence — Sample size calculations were based on the primary statistical analysis (see above); Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.2 to 2.6] — Hazard ratio was adjusted for age, BMI, smoking, and treated hypertension

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected over a period of 4 years.
Description: All study participants were asked for adverse events at each follow-up.
Arm/Group | NuvaRing | Combined Oral Contraceptives (COC)
Serious Adverse Events (participants affected / at risk) | 577/17084 | 751/17016
Other Adverse Events (participants affected / at risk) | 0/16864 | 0/16431
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NuvaRing (N=17084) | Combined Oral Contraceptives (COC) (N=17016)
Infectious diseases (Infections and infestations) | 20 | 30
Neoplasms, malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 19
Neoplasms, benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 10
Diseases of the blood and blood-forming organs (Blood and lymphatic system disorders) | 3 | 3
Endocrine diseases (Endocrine disorders) | 7 | 8
Psychiatric & neurological disorders (Psychiatric disorders) | 42 | 52
Eye (Eye disorders) | 3 | 5
Ear (Ear and labyrinth disorders) | 8 | 9
Cardiovascular system (Cardiac disorders) | 53 | 75
Respiratory system (Respiratory, thoracic and mediastinal disorders) | 40 | 54
Digestive system (Gastrointestinal disorders) | 126 | 169
Skin (Skin and subcutaneous tissue disorders) | 19 | 22
Muscosceletal system & connective tissue (Musculoskeletal and connective tissue disorders) | 19 | 26
Genitourinary system (Reproductive system and breast disorders) | 112 | 144
Injury, poisening, accidents, etc (Injury, poisoning and procedural complications) | 102 | 125

LIMITATIONS AND CAVEATS:
In non-experimental studies the possibility of bias and residual confounding can never be entirely eliminated. The findings may exclude large, but not small relative risks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No